CLINICAL TRIAL: NCT04907526
Title: Phase I Study of Intramyocardial Injection of Autologous Umbilical Cord Blood-Derived Mononuclear Cells During Fontan Surgical Palliation of Single Right Ventricle-Dependent Congenital Heart Disease
Brief Title: Intramyocardial Injection of Autologous UCB-MNC During Fontan Surgery for SRV Dependent CHD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy J Nelson, MD, PhD (Other)
Collaborators: Mayo Clinic (Other); University of Oklahoma (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Los Angeles (Other); Children's Hospitals and Clinics of Minnesota (Other); Children's Hospital Colorado (Other); Ochsner Health System (Other); Children's of Alabama (Other); Children's Hospital Medical Center, Cincinnati (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor-Investigator, Timothy J Nelson, MD, PhD, Program Director, ReGen Theranostics, Inc.
Organization: ReGen Theranostics, Inc. (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-000088
Record Dates: First submitted 2021-05-12; First posted 2021-05-28 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease, SRV Dependent
Keywords: Hypoplastic Left Heart Syndrome; HLHS; Congenital Heart Disease; Umbilical Cord Blood; UCB; Cord Blood; Stem Cells; Regenerative therapy; Stage III Fontan; Fontan surgery
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Autologous (self) mononuclear cells derived from umbilical cord blood and that meet all release criteria are injected into the surface of the right heart muscle to achieve the target dose of 3 million cells per kilogram of body weight. This is a one time treatment at the time of Stage III Fontan surgery.
  Interventions: Biological: Autologous mononuclear cells
- Control Arm (No Intervention): Control cohort not receiving the cell product, which will be enrolled and followed using the same inclusion/exclusion criteria and follow-up requirements as the treatment arm.

INTERVENTIONS:
Biological: Autologous mononuclear cells — Autologous mononuclear cells delivered into right ventricle at time of Stage III Fontan surgery.
  Arms: Treatment Arm

SUMMARY:
Researchers want to better understand what happens to the heart when the autologous (from one's own body) stem cells are injected directly into muscle of the right side of the heart during the Fontan (Stage III) surgery. They want to see if there are changes in the electrical activity, the structure, and the function of the heart following this stem cell-based therapy. Researchers will compare the results from people who receive the stem cells to the results from people who do not receive the stem cells.

DETAILED DESCRIPTION:
This Phase I study is a multicenter, prospective, open-label, non-randomized study designed to evaluate the safety, of autologous UCB-MNC delivered into the right ventricular myocardium of subjects with severe CHD defined by single right ventricular dependent circulatory systems at the time of a planned Fontan surgical palliation. This will be achieved by comparing the data collected in the treatment arm to the equivalent data collected in the control arm. The purpose of this non-randomized open-label Phase I clinical study is to prospectively evaluate the safety, as measured by the short-term and long-term safety endpoints and change in baseline comparatives, for the autologous UCB-MNC intramyocardial injections into the single, morphologically right ventricle of subjects with severe CHD requiring Fontan surgical palliation. The treatment group will be compared to an untreated control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a congenital hear defect with functionally single right ventricle (such as HLHS, HLHS variants, unbalanced AV septal defect with R dominance, DORV with Hypoplastic LV) undergoing Fontan surgical palliation
* At least 2 and less than or equal to 5 years of age at time of Fontan surgical palliation
* For subjects enrolling in the treatment arm, previous participation in clinical trial Umbilical Cord Blood Collection and Processing for Hypoplastic Left Heart Syndrome patients (NCT01856049) with autologous UCB-MNC product collected and available for distribution is required.

Exclusion Criteria:

* History of DMSO reaction (treatment arm only subjects).
* Parent(s) or legal guardian unwilling to have their child participate or unwilling to follow the study procedures.
* Severe chronic diseases at the discretion of the treating physician.
* Extensive extra-cardiac syndromic features.
* History of cancer.
* Any of the following complications of his/her congenital heart disease:

  * any condition requiring urgent, or unplanned intervention procedure within 15 days prior to Fontan surgical palliation, unless complete and full cardiac recovery is documented by site investigator.
  * severe pulmonary hypertension (reported in the medical record as >70% systemic pressure)
  * Other clinical concerns as documented by a site investigator that would predict (more likely to happen than not to happen) a risk of severe complications or very poor outcome, not directly related tot he stem cell product or its injection procedure, during or after Fontan surgical palliation.
* Individuals with severe heart failure that requires heart transplantation
* Individuals with refractory or worsening arrhythmia
* Individuals with an automated implantable cardioverter defibrillator (AICD) or pacemaker
* Patient with prior surgical complications during the Fontan surgical palliation that resulted in or could be reasonably expected to significantly decrease cardiac function

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Short-term safety | Within 3 months post Fontan surgery
  Measure of new or worsening adverse events

SECONDARY OUTCOMES:
Long term safety | Within 2 years post Fontan surgery
  Measure of new or worsening adverse events
Right ventricular function | Baseline, hospital discharge (up to 30 days post Fontan surgery), 3 months post Fontan surgery
  Change from baseline Transthoracic Echocardiogram right ventricular function as measured by biplane Fractional Area Change (FAC) at discharge and 3 months
High sensitivity Troponin T | 3 hours post enrollment, 6 hours post enrollment, hospital discharge (up to 30 days post Fontan surgery)
  Change from baseline in High sensitivity Troponin T at 3 hours and 6 hours after enrollment and at hospital discharge
NT-pro-BNP | Baseline, hospital discharge (up to 30 days post Fontan surgery), 3 months post Fontan surgery
  Change from baseline in NT-pro-BNP levels compared to baseline, at hospital discharge and at 3 months post-Fontan surgery
Panel Reactive Antibody | Baseline, hospital discharge (up to 30 days post Fontan surgery), 3 months post Fontan surgery
  Change from baseline in PRA levels at discharge and 3 months post-Fontan surgery compared to baseline.
Weight | Baseline, 3 months post-Fontan surgery, 12 months post-Fontan surgery
  Change from baseline in weight at 3 and 12 months post-Fontan surgery.
Cumulative days hospitalization | 3 months post discharge, 12 months post discharge
  Cumulative days of hospitalization per patient at 3 and 12 months post-Fontan surgery discharge
PROMIS Parent Proxy Scale v1.0-Global Health 7 | Baseline, hospital discharge (up to 30 days post Fontan surgery), 3 months, 12 months, 18 months, 24 months
  Change from baseline in PROMIS Parent Proxy Scale v1.0-Global Health 7 at discharge, 3, 12, 18, and 24 months post-Fontan surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Dearani, Principal Investigator — Mayo Clinic; Harold M Burkhart, Principal Investigator — Children's Hospital Oklahoma University Medical Center; Joseph w Rossano, Principal Investigator — Children's Hospital of Philadelphia; David M Overman, Principal Investigator — Children's Minnesota; John D Cleveland, MD, Principal Investigator — Children's Hospital Los Angeles; James Jaggers, MD, Principal Investigator — Children's Hospital Colorado; Benjamin Peeler, MD, Principal Investigator — Ochsner Health System; Waldemer Carlo, M.D., Principal Investigator — University of Alabama at Birmingham; James Tweddell, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Jason Maynes, MD, Principal Investigator — The Hospital forSick Children
Locations (6):
- United States (6):
  - University of Alabama Medical Center, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No